CLINICAL TRIAL: NCT00000899
Title: Effect of Cytoreductive Chemotherapy Combined With Highly Active Antiretroviral Therapy on Lymph Node HIV DNA in HIV-Infected Subjects
Brief Title: A Study on the Effect of Chemotherapy Combined With Anti-HIV Drugs in HIV-Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 380; 11341 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Cyclophosphamide; Dose-Response Relationship, Drug; Drug Therapy, Combination; Granulocyte Colony-Stimulating Factor; Combined Modality Therapy; Antineoplastic Agents; Lymph Nodes; Stavudine; HIV Protease Inhibitors; Lamivudine; DNA, Viral; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Nelfinavir; Antineoplastic Agents, Alkylating
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; Lamivudine; Filgrastim; Stavudine; Cyclophosphamide

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Filgrastim
Drug: Stavudine
Drug: Cyclophosphamide

SUMMARY:
The purpose of this study is to determine the safety of anti-HIV drugs combined with low-dose chemotherapy (consisting of cyclophosphamide [CTX]) in HIV-positive patients. This study examines whether this combination therapy can reduce the number of HIV-infected cells hidden in the lymph nodes and blood.

Current anti-HIV drug treatments can greatly reduce the levels of HIV in the human body. However, HIV can hide in certain immune cells and escape the drugs' effects. Chemotherapy using CTX destroys these immune cells. When used with standard anti-HIV drug treatments, CTX may be able to speed up the elimination of HIV-infected cells.

DETAILED DESCRIPTION:
HAART is a potent suppressor of plasma and lymph node HIV RNA. However, studies suggest that HAART cannot significantly diminish reservoirs of chronically HIV-infected cells. Strategies designed to eradicate all HIV infection should seek to actively target these reservoirs. CTX administration has been shown to eliminate a large number of lymphoid tissue T cells and macrophages, appearing to actively target chronically HIV-infected cells. As lymphoid organs are repopulated following initial depletion with CTX, HAART may protect repopulating cells from becoming HIV-infected, resulting in a net additional removal of the HIV-infected lymphoid reservoir.

In Step 1 of this 2-step protocol, all patients receive a HAART regimen of nelfinavir (NFV) plus stavudine (d4T) plus lamivudine (3TC). Patients who achieve an acceptable virologic response, defined as 2 consecutive HIV RNA determinations below 500 copies/ml at least 2 weeks apart between Weeks 4 and 16 of Step 1 [AS PER AMENDMENT 10/30/98: defined as 2 consecutive plasma HIV RNA determinations below 50 copies/ml by the Roche Ultrasensitive assay within a 4-week period between Weeks 4 and 24], are randomized to Arm A or B of Step 2. In Arm A, patients receive NFV plus d4T plus 3TC. In Arm B, patients receive NFV plus d4T plus 3TC plus 3 escalating doses of CTX at 6-week intervals. Patients in both arms are followed for at least 52 weeks following randomization to Step 2. During this time, patients undergo blood tests and lymph node biopsies to measure HIV DNA and RNA levels and to characterize the T cell population. Additionally, patients undergo a chest CT of the thymus before randomization to Step 2 and at Week 52 of Step 2. Cerebrospinal fluid may be obtained at Week 52 to determine the amount of HIV RNA and DNA present. [AS PER AMENDMENT 10/30/98: G-CSF is given after the first dose of CTX, at the discretion of the investigator, and after the second and third doses, for up to 14 days, until the absolute neutrophil count is 10,000 cells/mm3. Also, CTX doses may be modified based on pharmacokinetic study results.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 count above 300 cells/mm3 within 30 days of study entry.
* Have an HIV viral load between 10,000 and 200,000 copies/ml.
* Are between the ages of 18 and 50.
* Agree to practice abstinence or to use a barrier method of birth control during the study (such as condoms).

Exclusion Criteria

You may not be eligible for this study if you:

* Have had cancer requiring chemotherapy or radiotherapy or certain nervous system diseases.
* Are sensitive to E. coli-derived proteins.
* Have an active AIDS-defining illness.
* Require certain medications.
* Are pregnant or breast-feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Bartlett, MD, Study Chair — Duke Univ Med Ctr
Locations (2):
- United States (2):
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] Bartlett JA, Silberman M, Miralles GD, Sevin A, Pruitt S, Ottinger J, Gryszowka V, Fiscus S, Bucy BP. Antiretroviral therapy (ART) plus cyclophosphamide (CTX) to diminish HIV DNA in lymphoid tissue. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 16)
- [Background] Bartlett JA, Miralles GD, Sevin AD, Silberman M, Pruitt SK, Ottinger J, Gryszowska V, Fiscus SA, Bucy RP; ACTG 380 Study Team. Addition of cyclophosphamide to antiretroviral therapy does not diminish the cellular reservoir in HIV-infected persons. AIDS Res Hum Retroviruses. 2002 May 20;18(8):535-43. doi: 10.1089/088922202753747888. PMID 12036483